CLINICAL TRIAL: NCT01476306
Title: Providing Specialty Care to Individuals With Parkinsonism Directly in Their Homes Via Web-based Video Conferencing- A Comparative Effectiveness Study
Acronym: TELEMED-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00044310
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Parkinson Disease
Keywords: feasibility; effectiveness; Parkinson disease care; care via telemedicine
MeSH Terms: conditions — Parkinson Disease | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-patient care (Placebo Comparator)
  Interventions: Other: Usual care
- Telemedicine care (Experimental)
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Patient will receive care using HIPAA-compliant web-based videoconferencing rather than their usual in-patient care.
  Arms: Telemedicine care
Other: Usual care — Patients in this group will receive care as they usually do with the physician.
  Arms: In-patient care

SUMMARY:
The investigators will conduct a two-arm, parallel group, randomized comparative effectiveness study across two sites to increase specialty access and improve care for individuals with Parkinsonism and their caregivers. Twenty individuals with Parkinsonism will be recruited from Johns Hopkins University and the University of Rochester (approximately ten from each site). They will then be randomized to either continue their usual in-person care with a specialist or to receive care with their specialist via telemedicine in their home. Following an in-person baseline/screening visit, approximately ten individuals in the first arm (virtual house calls) will receive three visits with a movement disorder specialist via telemedicine (using web-based video conferencing) in their home. Approximately ten individuals in the second (control) arm will receive three in-person visits at an academic medical center with the same specialists. Approximately two weeks after the completion of each clinical visit, a nurse or coordinator will call the patient to call to address any questions or ensure appropriate understanding of the recommendation (for both telemedicine and control arms). Overall, the study - consistent with a national priority for comparative effectiveness research - will compare the use of telemedicine to manage Parkinsonism to usual care.

DETAILED DESCRIPTION:
1. Abstract

   The research's overall objective is to improve care for individuals with Parkinsonism. Parkinsonism is clinically determined as the presence of at least 2 of the following: 1) rest tremor, 2) bradykinesia, 3) cogwheel rigidity, or 4) difficulty with gait or balance. The most common cause of Parkinsonism is Parkinson disease. Parkinson disease is a chronic condition whose burden is growing both in the United States and globally. However, access to specialty care is limited chiefly to urban areas and is frequently inefficient. One way to remove geographic barriers to care is through the use of web-based video conferencing (telemedicine).

   To evaluate the study's aims, the investigators will conduct a seven-month randomized controlled study of twenty patients with Parkinsonism across two sites to contrast the comparative effectiveness of standard in-person specialty visits versus those conducted via web-based video conferencing (telemedicine). It is hypothesized that these "virtual house calls" will be feasible, clinically non-inferior to usual care, and economically valuable. This research will expand the geographic scope of specialty care and provide a national model for providing home-based, patient-centered, cost-effective care to those with Parkinsonism anywhere they live.
2. Objectives (include all primary and secondary objectives)

The specific objectives of the study are as follows:

Aim 1: To evaluate the feasibility of providing specialty care to individuals with Parkinsonism via web-based video conferencing (telemedicine) in their homes by calculating the proportion of specialty visits completed as scheduled.

Hypothesis 1: Individuals receiving care via telemedicine in their homes will complete at least 80% of their visits as scheduled.

Aim 2: To explore the clinical benefits, as measured by the change from baseline in quality of life as measured by the Parkinson Disease Questionnaire 39 (PDQ-39).

Hypothesis 2: In this pilot study, the change in quality of life will be comparable between the two groups.

Aim 3: To explore the economic benefit of providing specialty care via telemedicine in the home.

Hypothesis 3: For patients and caregivers, travel and labor savings from receiving care in the home will outweigh technology costs for telemedicine visits.

ELIGIBILITY:
Inclusion Criteria:

* The principal eligibility criteria for participants are the following: age greater than 30, clinical diagnosis of idiopathic Parkinsonism, ability to converse in English, ability and willingness to provide informed consent and complete study requirements, and access to a computer with broadband internet.

Exclusion Criteria:

* The main exclusion criterion is a condition (e.g., prominent psychosis) that in the investigator's judgment would preclude participation in a telemedicine visit. Participants may identify a principal caregiver for optional participation in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Feasibility | 7 months
  Percentage of visits completed as scheduled, number of individuals in telemedicine arm who require in-person visit, number of in-person visits required by individuals in telemedicine arm, proportion of completed telemedicine visits versus in-person visits

SECONDARY OUTCOMES:
Clinical Benefits | 7 months
  Unified Parkinson Disease Ration Scale (UPDRS) part III, Montreal Cognitive Assessment (MoCA), Hoehn and Yahr, Patient Assessment of Care for Chronic Conditions (PACIC) Survey, Patient satisfaction
Economic impact | 7 months
  Travel, time, facilities fees

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medical Institutes, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Dorsey ER, Venkataraman V, Grana MJ, Bull MT, George BP, Boyd CM, Beck CA, Rajan B, Seidmann A, Biglan KM. Randomized controlled clinical trial of "virtual house calls" for Parkinson disease. JAMA Neurol. 2013 May;70(5):565-70. doi: 10.1001/jamaneurol.2013.123. PMID 23479138